CLINICAL TRIAL: NCT00647556
Title: A Comparative Study of Adapalene Gel 0.3% Versus Tretinoin 0.05% Emollient Cream, for the Treatment of Photodamage
Brief Title: Adapalene Gel 0.3% Versus Tretinoin 0.05% Emollient Cream for Treatment of Photodamage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US10067
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Results first posted 2011-02-24 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2012-09

CONDITIONS: Photoaging
MeSH Terms: interventions — Adapalene; Gels; Tretinoin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- adapalene (Active Comparator): adapalene
  Interventions: Drug: adapalene gel, 0.3%
- tretinoin (Active Comparator): Tretinoin
  Interventions: Drug: tretinoin 0.05% emollient cream

INTERVENTIONS:
Drug: adapalene gel, 0.3% — applied topically once daily in the evening
  Other Names: Differin® 0.3% Gel
  Arms: adapalene
Drug: tretinoin 0.05% emollient cream — applied topically once daily in the evening
  Other Names: tretinoin emollient cream 0.05%
  Arms: tretinoin

SUMMARY:
The primary purpose of this study is to compare the efficacy of adapalene (Differin®) gel 0.3% and tretinoin 0.05% emollient cream for the treatment of signs of photodamage, with tolerability assessment as a secondary objective.

DETAILED DESCRIPTION:
Same as above.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 40 years of age and older with Fitzpatrick skin types I through III
* Clinically moderate to severe photodamage

Exclusion Criteria:

* Subjects with history of laser resurfacing, dermabrasion, medium or deep chemical peel of the face
* Subjects with diagnosis of skin cancer within 3 months of study entry
* Subjects who have had superficial chemical peels, exfoliation or microdermabrasion of the face within 3 months of study entry
* Subjects who have had botulinum toxin for facial rejuvenation within 6 months of study entry and are unwilling to refrain from botulinum toxin treatments during the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: First subject was enrolled on June 17, 2008 and the last subject was enrolled on July 24, 2009.
Pre-assignment Details: Wash-out period at baseline: 2 wks topical alpha-hydroxy, glycolic, salicylic, lactic, & beta-hydroxy acids, topical vitamin A, ascorbic acid, vitamin E, corticosteroids on face; 4 wks systemic corticosteroids; 3 mos topical retinoids, superficial chemical peels/exfoliation/microdermabrasion; 6 mos botulinum toxin on the face; 1 yr oral retinoids.
Groups:
- Differin® Gel, 0.3%: adapalene gel 0.3% - apply once daily in the evening for 24 weeks
- Tretinoin Emollient Cream: Tretinoin Emollient Cream 0.05% - apply topically once daily in the evening for 24 weeks
Period: Overall Study
Arm/Group | Differin® Gel, 0.3% | Tretinoin Emollient Cream
Started | 15 | 15
Completed | 12 | 13
Not Completed | 3 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Surgery for pre-existing neck pain | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Differin® Gel, 0.3% | Tretinoin Emollient Cream | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (11.37) | 61.3 (9.58) | 61.1 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Overall Integrated Assessment of Photodamage at Week 24
Description: Number of participants who improved (a decrease by at least one point) in Overall Integrated Assessment of Photodamage from baseline to week 24. Overall Integrated Assessment of Photodamage is a scale from 0 - 5 (0 = None, 1 = Minimal, 2 = Mild, 3 - Moderate, 4 = Severe and 5 = Very Severe) with 0 being best and 5 being worst.
Time Frame: baseline to week 24
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Differin® Gel, 0.3% | Tretinoin Emollient Cream
Number analyzed (Participants) | 15 | 15
participants | 6 | 10

2. Secondary Outcome: Photonumeric Scale for the Assessment of Photodamage From Baseline to Week 12 and Baseline to Week 24
Description: Number of participants in each category of the Photonumeric Scale for the Assessment of Photodamage from baseline to week 12 and baseline to week 24. Photonumeric Scale consisted of 9 categories (Fine Wrinkling, Mottled Pigmentation, Irregular Depigmentation, Lentigines, Coarse Wrinkling, Elastosis, Tactile Roughness, Telangiectasia, and Actinic Keratosis. These were evaluated on a scale from 0 - 4 (0 = None, 1 = Minimal, 2 = Mild, 3 = Moderate and 4 = Severe) with 0 being best and 4 being worst.
Time Frame: baseline, week 12 and week 24
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Differin® Gel, 0.3% | Tretinoin Emollient Cream
Number analyzed (Participants) | 15 | 15
participants
  Fine wrinkling baseline None (0) | 0 | 0
  Fine wrinkling baseline Minimal (1) | 0 | 0
  Fine wrinkling baseline Mild (2) | 3 | 2
  Fine wrinkling baseline Moderate (3) | 12 | 11
  Fine wrinkling baseline Severe (4) | 0 | 2
  Fine wrinkling week 12 None (0) | 0 | 0
  Fine wrinkling week 12 Minimal (1) | 1 | 1
  Fine wrinkling week 12 Mild (2) | 9 | 4
  Fine wrinkling week 12 Moderate (3) | 5 | 9
  Fine wrinkling week 12 Severe (4) | 0 | 1
  Fine wrinkling week 24 None (0) | 0 | 1
  Fine wrinkling week 24 Minimal (1) | 2 | 2
  Fine wrinkling week 24 Mild (2) | 8 | 4
  Fine wrinkling week 24 Moderate (3) | 5 | 7
  Fine wrinkling week 24 Severe (4) | 0 | 1
  Mottled pigmentation baseline None (0) | 0 | 0
  Mottled pigmentation baseline Minimal (1) | 0 | 4
  Mottled pigmentation baseline Mild (2) | 7 | 8
  Mottled pigmentation baseline Moderate (3) | 8 | 2
  Mottled pigmentation baseline Severe (4) | 0 | 1
  Mottled pigmentation week 12 None (0) | 0 | 0
  Mottled pigmentation week 12 Minimal (1) | 1 | 7
  Mottled pigmentation week 12 Mild (2) | 7 | 5
  Mottled pigmentation week 12 Moderate (3) | 6 | 3
  Mottled pigmentation week 12 Severe (4) | 1 | 0
  Mottled pigmentation week 24 None (0) | 1 | 0
  Mottled pigmentation week 24 Minimal (1) | 3 | 10
  Mottled pigmentation week 24 Mild (2) | 6 | 4
  Mottled pigmentation week 24 Moderate (3) | 4 | 1
  Mottled pigmentation week 24 Severe (4) | 1 | 0
  Irregular depigmentation baseline None (0) | 1 | 1
  Irregular depigmentation baseline Minimal (1) | 5 | 7
  Irregular depigmentation baseline Mild (2) | 6 | 5
  Irregular depigmentation baseline Moderate (3) | 3 | 2
  Irregular depigmentation baseline Severe (4) | 0 | 0
  Irregular depigmentation week 12 None (0) | 1 | 1
  Irregular depigmentation week 12 Minimal (1) | 6 | 9
  Irregular depigmentation week 12 Mild (2) | 6 | 4
  Irregular depigmentation week 12 Moderate (3) | 2 | 1
  Irregular depigmentation week 12 Severe (4) | 0 | 0
  Irregular depigmentation week 24 None (0) | 1 | 1
  Irregular depigmentation week 24 Minimal (1) | 7 | 9
  Irregular depigmentation week 24 Mild (2) | 5 | 5
  Irregular depigmentation week 24 Moderate (3) | 2 | 0
  Irregular depigmentation week 24 Severe (4) | 0 | 0
  Lentigines baseline None (0) | 0 | 0
  Lentigines baseline Minimal (1) | 2 | 3
  Lentigines baseline Mild (2) | 5 | 9
  Lentigines baseline Moderate (3) | 7 | 2
  Lentigines baseline Severe (4) | 1 | 1
  Lentigines week 12 None (0) | 0 | 0
  Lentigines week 12 Minimal (1) | 3 | 5
  Lentigines week 12 Mild (2) | 7 | 9
  Lentigines week 12 Moderate (3) | 5 | 1
  Lentigines week 12 Severe (4) | 0 | 0
  Lentigines week 24 None (0) | 1 | 0
  Lentigines week 24 Minimal (1) | 3 | 7
  Lentigines week 24 Mild (2) | 7 | 7
  Lentigines week 24 Moderate (3) | 4 | 1
  Lentigines week 24 Severe (4) | 0 | 0
  Coarse wrinkling baseline None (0) | 0 | 0
  Coarse wrinkling baseline Minimal (1) | 1 | 0
  Coarse wrinkling baseline Mild (2) | 10 | 5
  Coarse wrinkling baseline Moderate (3) | 2 | 7
  Coarse wrinkling baseline Severe (4) | 2 | 3
  Coarse wrinkling week 12 None (0) | 0 | 0
  Coarse wrinkling week 12 Minimal (1) | 2 | 0
  Coarse wrinkling week 12 Mild (2) | 9 | 8
  Coarse wrinkling week 12 Moderate (3) | 2 | 4
  Coarse wrinkling week 12 Severe (4) | 2 | 3
  Coarse wrinkling week 24 None (0) | 0 | 0
  Coarse wrinkling week 24 Minimal (1) | 2 | 2
  Coarse wrinkling week 24 Mild (2) | 8 | 6
  Coarse wrinkling week 24 Moderate (3) | 3 | 4
  Coarse wrinkling week 24 Severe (4) | 2 | 3
  Elastosis baseline None (0) | 0 | 0
  Elastosis baseline Minimal (1) | 1 | 1
  Elastosis baseline Mild (2) | 7 | 5
  Elastosis baseline Moderate (3) | 6 | 8
  Elastosis baseline Severe (4) | 1 | 1
  Elastosis week 12 None (0) | 0 | 0
  Elastosis week 12 Minimal (1) | 1 | 1
  Elastosis week 12 Mild (2) | 9 | 6
  Elastosis week 12 Moderate (3) | 4 | 7
  Elastosis week 12 Severe (4) | 1 | 1
  Elastosis week 24 None (0) | 0 | 0
  Elastosis week 24 Minimal (1) | 2 | 3
  Elastosis week 24 Mild (2) | 10 | 8
  Elastosis week 24 Moderate (3) | 3 | 3
  Elastosis week 24 Severe (4) | 0 | 1
  Tactile Roughness baseline None (0) | 0 | 1
  Tactile Roughness baseline Minimal (1) | 7 | 4
  Tactile Roughness baseline Mild (2) | 3 | 7
  Tactile Roughness baseline Moderate (3) | 4 | 3
  Tactile Roughness baseline Severe (4) | 1 | 0
  Tactile Roughness week 12 None (0) | 0 | 1
  Tactile Roughness week 12 Minimal (1) | 9 | 6
  Tactile Roughness week 12 Mild (2) | 5 | 7
  Tactile Roughness week 12 Moderate (3) | 0 | 0
  Tactile Roughness week 12 Severe (4) | 1 | 1
  Tactile Roughness week 24 None (0) | 0 | 1
  Tactile Roughness week 24 Minimal (1) | 10 | 11
  Tactile Roughness week 24 Mild (2) | 4 | 3
  Tactile Roughness week 24 Moderate (3) | 0 | 0
  Tactile Roughness week 24 Severe (4) | 1 | 0
  Telangiectasia baseline None (0) | 0 | 0
  Telangiectasia baseline Minimal (1) | 0 | 4
  Telangiectasia baseline Mild (2) | 6 | 5
  Telangiectasia baseline Moderate (3) | 9 | 4
  Telangiectasia baseline Severe (4) | 0 | 2
  Telangiectasia week 12 None (0) | 0 | 0
  Telangiectasia week 12 Minimal (1) | 2 | 4
  Telangiectasia week 12 Mild (2) | 4 | 5
  Telangiectasia week 12 Moderate (3) | 8 | 5
  Telangiectasia week 12 Severe (4) | 1 | 1
  Telangiectasia week 24 None (0) | 0 | 0
  Telangiectasia week 24 Minimal (1) | 3 | 5
  Telangiectasia week 24 Mild (2) | 4 | 3
  Telangiectasia week 24 Moderate (3) | 7 | 6
  Telangiectasia week 24 Severe (4) | 1 | 1
  Actinic keratosis baseline None (0) | 8 | 9
  Actinic keratosis baseline Minimal (1) | 5 | 3
  Actinic keratosis baseline Mild (2) | 1 | 1
  Actinic keratosis baseline Moderate (3) | 1 | 2
  Actinic keratosis baseline Severe (4) | 0 | 0
  Actinic keratosis week 12 None (0) | 9 | 9
  Actinic keratosis week 12 Minimal (1) | 5 | 4
  Actinic keratosis week 12 Mild (2) | 0 | 2
  Actinic keratosis week 12 Moderate (3) | 0 | 0
  Actinic keratosis week 12 Severe (4) | 1 | 0
  Actinic keratosis week 24 None (0) | 12 | 8
  Actinic keratosis week 24 Minimal (1) | 2 | 5
  Actinic keratosis week 24 Mild (2) | 0 | 2
  Actinic keratosis week 24 Moderate (3) | 0 | 0
  Actinic keratosis week 24 Severe (4) | 1 | 0

3. Secondary Outcome: Number of Participants Who Improved (a Decrease of at Least One Point) in Overall Integrated Assessment of Photodamage From Baseline to Week 12.
Description: Number of participants who improved in Overall Integrated Assessment of Photodamage from baseline to week 12. Overall Integrated Assessment of Photodamage was evaluated on a scale from 0 - 5 (0 = None, 1 = Minimal, 2 = Mild, 3 = Moderate 4 = Severe and 5 = Very Severe) with 0 being best and 5 being worst.
Time Frame: baseline to week 12
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Differin® Gel, 0.3% | Tretinoin Emollient Cream
Number analyzed (Participants) | 15 | 15
participants | 6 | 4

4. Secondary Outcome: Number of Participants in Each Category of the Subject Evaluation of Improvement at Week 12 and Week 24
Description: Number of participants in each category of the Subject Evaluation of Improvement at week 12 and week 24. Subject Evaluation of Improvement was evaluated on a scale from 0 - 6 (0 = Complete Improvement, 1 = Almost (~90%) Improvement, 2 = Marked (~75%) Improvement, 3 = Moderate (~50%) Improvement, 4 = Slight (~25%) Improvement, 5 = No Change, 6 = Worse) with 0 being best and 6 being worst.
Time Frame: week 12 and week 24
Population: ITT (Intent to Treat; LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Differin® Gel, 0.3% | Tretinoin Emollient Cream
Number analyzed (Participants) | 15 | 15
participants
  week 12 Complete Improvement | 0 | 0
  week 12 Almost Complete Improvement | 0 | 0
  week 12 Marked Improvement | 4 | 2
  week 12 Moderate Improvement | 4 | 5
  week 12 Slight Improvement | 4 | 4
  week 12 No Change | 0 | 2
  week 12 Worse | 0 | 0
  week 12 Missing | 3 | 2
  week 24 Complete Improvement | 0 | 0
  week 24 Almost Complete Improvement | 3 | 1
  week 24 Marked Improvement | 2 | 4
  week 24 Moderate Improvement | 4 | 4
  week 24 Slight Improvement | 3 | 1
  week 24 No Change | 0 | 5
  week 24 Worse | 0 | 0
  week 24 Missing | 3 | 0

5. Secondary Outcome: Number of Participants in Each Category of the Investigator Evaluation of Global Response (Improvement) at Week 12 and Week 24
Description: Number of participants in each category of the Investigator Evaluation of Global Response (Improvement) at week 12 and week 24. Investigator Evaluation of Global Response (Improvement) is evaluated on a scale from 0 - 6 (0 = Complete Response, 1 = Almost Complete (~90%) Response, 2 = Marked (~75%) Response, 3 = Moderate (~50%) Response, 4 = Slight (~25%) Response, 5 = No Response and 6 = Worsening) with 0 being best and 6 being worst.
Time Frame: week 12 and week 24
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Differin® Gel, 0.3% | Tretinoin Emollient Cream
Number analyzed (Participants) | 15 | 15
participants
  week 12 Complete Response | 0 | 0
  week 12 Almost Complete Response | 0 | 0
  week 12 Marked Response | 0 | 1
  week 12 Moderate Response | 2 | 4
  week 12 Slight Response | 9 | 6
  week 12 No Response | 1 | 2
  week 12 Worsening | 0 | 0
  week 12 Missing | 3 | 2
  week 24 Complete Response | 0 | 0
  week 24 Almost Complete Response | 0 | 0
  week 24 Marked Response | 2 | 0
  week 24 Moderate Response | 2 | 8
  week 24 Slight Response | 6 | 4
  week 24 No Response | 2 | 3
  week 24 Worsening | 0 | 0
  week 24 Missing | 3 | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Subjects were asked if there had been any change in their health at each study visit; information obtained was recorded as adverse event(s), when applicable.
Arm/Group | Differin® Gel, 0.3% | Tretinoin Emollient Cream
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 7/15 | 14/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Differin® Gel, 0.3% (N=15) | Tretinoin Emollient Cream (N=15)
Application site bleeding (General disorders) | 0 (0) | 1 (1)
Application site burn (General disorders) | 1 (2) | 0 (0)
Application site dermatitis (General disorders) | 0 (0) | 2 (3)
Application site irritation (General disorders) | 1 (1) | 0 (0)
Application site reaction (General disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Chlamydial infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gonorrhea (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 2 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Open wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Terminal dribbling (Renal and urinary disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator has the right to publish or present the data resulting from this study, with agreed upon reviews by all interested parties, and in accordance with any confidentiality agreements that may exist.